CLINICAL TRIAL: NCT06195527
Title: PEMBRO-K : Evaluation of Pembrolizumab Therapeutic Pharmacological Monitoring Benefit in Non-small Cell Bronchopulmonary Cancer (NSCLC)
Brief Title: PEMBRO-K : Evaluation of Pembrolizumab Therapeutic Pharmacological Monitoring Benefit in NSCLC
Acronym: PEMBRO-K
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Other Study IDs: 49RC21_0253; 2023-A02527-38 (Other: n° IdRCB)
Record Dates: First submitted 2023-12-22; First posted 2024-01-08 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Solid cancers and their therapeutic management remain a major public health problem due to their increasing prevalence and associated mortality. Among solid cancers, lung cancer ranks 4th among incident cancers. The prognosis remains poor, 33,117 deaths were recorded in France in 2018. Two histological forms of bronchopulmonary cancer are distinguished: non-small cell lung cancers (NSCLC), which represent 85% of bronchopulmonary cancer, and small cell lung cancers. The most common forms of NSCLC are adenocarcinoma, squamous cell carcinoma and large cell carcinoma.

The emergence of new so-called targeted therapies has considerably modified the management and prognosis of oncology patients and in particular of patients with NSCLC. These new molecules were developed following the molecular characterization of tumors on the one hand and on the other hand the characterization of the role of immunity in anti-tumor defense, particularly the Programmed Death receptor pathway 1 (PD-1). Blocking this pathway restores the anti-tumor potential of these lymphocytes. Pembrolizumab is a humanized monoclonal antibody that binds to the PD-1 receptor and blocks its interaction with the Programmed Death Ligand-1 (PDL1) and Programmed Death Ligand-2 (PDL2), expressed by tumor cells but also by cells in the microenvironment. tumor and by antigen-presenting cells. Pembrolizumab thus potentiates T cell responses, including anti-tumor responses, by blocking the binding of PD-1 with PDL1 and PDL2.

Pembrolizumab currently has marketing authorization (MA) for the treatment of NSCLC. Despite therapeutic progress due, among other things, to the emergence of anti-PD-1 antibodies including pembrolizumab, the prognosis of NSCLC remains poor and the use of pembrolizumab is sometimes limited by the occurrence of adverse effects.

The pharmacokinetics of pembrolizumab was studied pre-marketing in patients with melanoma, NSCLC or metastatic or unresectable carcinomas. However, there are no data relating to the pharmacokinetic (PK) / clinical response (pharmacodynamic / PD) relationship of pembrolizumab, in real life. No prospective pharmacological study has in fact been published to date, especially in patients treated as part of the management of NSCLC. The absence of such studies - in real life - constitutes a pitfall given the existence of a possible association between PK data and the clinical response and/or toxicity of pembrolizumab.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or more
* patient with NSCLC
* pembrolizumab treatment (monotherapy or not) with a placed line (peripheral catheter, PICC or implantable port)

Exclusion Criteria:

* objection to participate in the study
* patient under judicial protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a population pharmacokinetic study aimed at establishing the PK-PD relationship in patients with NSCLC treated with pembrolizumab (non-comparative descriptive study).
  Taking into account the half-life (26 days) and the time necessary to obtain the equilibrium state (16 weeks), the choice was made to take residual and peak samples during administrations. This sampling strategy will allow the construction and validation of the PK model.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2025-12-17 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Pembrolizumab efficiency Month 2 | month 2
  Pembrolizumab effectiveness according to RECIST's radiological criteria

SECONDARY OUTCOMES:
Pembrolizumab efficiency Month 4 | month 4
  Pembrolizumab effectiveness according to RECIST's radiological criteria
Pembrolizumab efficiency Month 12 | month 12
  Pembrolizumab effectiveness according to RECIST's radiological criteria
Pembrolizumab toxicity Month 18 | month 18
  All adverse/toxic reactions collected by Regional Safety center until 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume DREVIN, Doctor, Study Director — Angers University Hospital
Locations (2):
- France (2):
  - Angers University Hospital, Angers
  - CH Le Mans, Le Mans